CLINICAL TRIAL: NCT05213195
Title: NKG2D CAR-NK Cell Therapy in Patients With Refractory Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Professor, Zhejiang University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CARNK-002
Record Dates: First submitted 2021-12-25; First posted 2022-01-28 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Refractory Metastatic Colorectal Cancer
Keywords: Refractory Metastatic Colorectal Cancer; NKG2D; CAR-NK
MeSH Terms: conditions — Colorectal Neoplasms | interventions — NK Cell Lectin-Like Receptor Subfamily K; Automobiles; Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NKG2D CAR-NK (Experimental): NKG2D CAR-NK Cell Therapy in Patients With Refractory Metastatic Colorectal Cancer Will be intra-peritoneal infusion in Stage 1 and combined with intra-venous infusion in Stage 2. While in Stage 3, the investigators will expand to other cancer type at certain situation
  Interventions: Drug: NKG2D CAR-NK

INTERVENTIONS:
Drug: NKG2D CAR-NK — NKG2D CAR-NK infusion through peritoneal in stage 1 and later combined with intra venous in stage 2.
  Other Names: Natural killer group 2 member D (NKG2D) ligand-targeting chimeric antigen receptor (CAR) natural killer (NK) cells

SUMMARY:
NKG2D CAR-NK Cell Therapy in Patients With Refractory Metastatic Colorectal Cancer

DETAILED DESCRIPTION:
NKG2D CAR-NK Cell Therapy in Patients With Refractory Metastatic Colorectal Cancer Will be intra-peritoneal infusion in Stage 1 and combined with intra-venous infusion in Stage 2. While in Stage 3, the investigators will expand to other cancer type at certain situation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years (including boundary values), both male and female.
2. Patients with advanced colorectal cancer with abdominal metastasis who had previously failed standard therapy and no other feasible and effective treatment was available.
3. The expected survival period of the subject is ≥12 weeks.
4. Subjects should have at least one target lesion that can be assessed stably by CT or MRI according to RECIST V.1.1.

The target lesions had measurable diameter lines (tumor lesions with CT scan length ≥10 mm, lymph node lesions with CT scan short diameter ≥10 mm 15 mm, scanning layer thickness is no more than 5 mm). Or by laparoscopy, at least one of them had PCI scores Accurate, assessable target lesions.

5. ECOG physical status score is 0 ~ 1.

6. Subject has adequate organ and bone marrow function. Laboratory screening must meet the following criteria for all laboratory tests Results should be within the stable range described below and without continuous supportive treatment.

1. Blood test: WBC≥ 1.5×109/L; Platelet count PLT ≥60×109/L; Hemoglobin content Hb 8.0 g/dL or higher; Lymphocyte LYM≥0.4×109/L;
2. Blood biochemistry: serum creatinine ≤1.5 ×ULN, if serum creatinine > 1.5 ×ULN, creatinine clearance rate > 50mL/min (calculated according to the Cockcroft-Gault formula); Serum total bilirubin ≤1.5×ULN, ALT≤2 ×ULN, AST≤ 2 ×ULN (liver metastasis or liver cancer patients) ALT≤5 x ULN, AST≤5 x ULN).
3. Amylase and lipase ≤ 1.5 × ULN;
4. Routine urine examination: urinary protein < 2+.

   7. Left ventricular ejection fraction (LVEF) > 45% by color doppler echocardiography within one month

   8. Fertility status: Female patients of reproductive age or male patients with sexual partners of female patients of reproductive age are willing to sign informed consent,Use effective contraception from the beginning to 6 months after the last cell infusion (women of childbearing age include premenopausal women and postmenopausal women)

   Women within 2 years).

   9. Subject must sign and date written informed consent.

   10. Subjects must be willing and able to comply with scheduled treatment regimens, laboratory tests, follow-up visits, and other study requirements

   Exclusion Criteria:
   1. Pregnant and lactating women.
   2. Known history of human immunodeficiency virus (HIV) infection; Acute or chronic active hepatitis B (HBsAg positive);

   Acute or chronic active hepatitis C (positive for HCV antibody). Syphilis antibody positive; Epstein-barr virus DNA quantification

   500 copies; Cytomegalovirus (CMV) infection (IgM positive).

   3. Severe infection that is in the active stage or clinically poorly controlled.

   4. Existing heart disease requiring treatment or hypertension determined to be poorly controlled by the investigator (defined as standardized blood pressure reduction)

   Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure > 90 mmHg after treatment).

   5. Presence of any of the following cardiac clinical symptoms or diseases:

   A) Unstable angina pectoris;

   B) Myocardial infarction occurred within 1 year;

   C) Resting state ecg QTc > 450ms(male) or QTc > 470ms (female);

   D) Abnormalities of clinical significance (such as heart rate, conduction, morphological characteristics, etc.) detected by resting ecg examination

   Complete left bundle branch block or grade 3 heart block or grade 2 heart block or PR interval >

   250 ms;

   E) There are factors that increase the risk of prolonged QTc and abnormal heart rate, such as heart failure, hypokalemia, and congenital long QT

   Family history of long QT syndrome or sudden unexplained death of a direct family member under 40 years of age, or prolonged period of time

   Phase iii concomitant medication.

   6. Abnormal coagulation function (INR > 1.5× ULN), bleeding tendency or receiving thrombolytic or conventional anticoagulant therapy (e.g

   Warfarin or heparin) in patients requiring long-term antiplatelet therapy (aspirin > 300mg/day; Clopidogrel,

   Dose > 75mg/day).

   7. Subjects requiring systemic treatment with corticosteroids or other immunosuppressive agents during the treatment period.

   8. Blood oxygen saturation ≤95% (pulse oxygen test) before treatment.

   9. Received systemic steroids equivalent to > 15mg/ day of prednisone, excluding inhaled steroids, within 4 weeks prior to treatment.

   10. New arrhythmias, including but not limited to arrhythmias that could not be controlled by drugs, occurred in subjects prior to pretreatment with clear shower

   Often, low blood pressure requiring compression, bacterial, fungal, or viral infections requiring intravenous antibiotics. Use the test

   Subjects who received antibiotics to prevent infection were judged by the investigator to be eligible for further study.

   11. Known past or present hepatic encephalopathy requiring treatment; Patients who currently have or have a history of central nervous system disorders, such as epilepsy

   Seizures, cerebral ischemia/hemorrhage, dementia, cerebellar disease or any autoimmune disease associated with central nervous system involvement

   Disease; Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence of the patient's central nervous system

   General or meningeal metastases were not controlled and were deemed unsuitable for inclusion by the investigator.

   12. Patients with prior or concurrent malignancy, except for: Adequately treated basal cell or squamous cell carcinoma (adequate wound healing required prior to enrollment); Carcinoma in situ of cervical or breast cancer, treated curatively, with no signs of recurrence for at least 3 years prior to the study; The primary malignancy has been completely resected with complete remission for ≥5 years.

   13. Prior NK or CAR-NK immunotherapy.

   14. Received anti-PD-1 /PD-L1 monoclonal antibody treatment within 4 weeks prior to treatment.

   15. Subjects who have previously received other gene therapies.

   16. Subjects with severe mental disorders.

   17. Participated in other clinical studies in the past 1 month.

   18. The investigator assessed subjects' inability or unwillingness to comply with study protocol requirements.

   19. Subjects withdraw from the study for various reasons and cannot participate in the study again.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity#DLT# | 28 days
  Safety
Maximal Tolerable Dose#MTD# | 28 days
  tolerability evaluation

SECONDARY OUTCOMES:
Antitumor efficacy-Duration of response (DOR) | 52 weeks
  The period from the first evaluation of complete response ( CR) or partial response (PR) to the first evaluation of progressive disease (PD)or death of any cause.
Antitumor efficacy-Objective response rate (ORR) | 52 weeks
  The number of cases in which tumor size is reduced to partial response (PR) or complete response (CR) / the total number of evaluable cases (%).
Antitumor efficacy-Overall survival (OS) | 52 weeks
  The period from the first study treatment to any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No